CLINICAL TRIAL: NCT01991717
Title: An Open-label Investigator-masked Study Comparing Femtosecond Laser Assisted With Conventional Phacoemulsification Cataract Surgery
Brief Title: Victus Versus Conventional
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Matthias Bolz (Other)
Collaborators: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor-Investigator, Matthias Bolz, MD, Augenabteilung Allgemeines Krankenhaus Linz
Organization: Augenabteilung Allgemeines Krankenhaus Linz (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13A06
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Cataract
Keywords: Victus; lensfragmentation; femtosecond laser assisted; capsulotomy,; manual, continuous curvilinear capsulorhexis (CCC); effective phaco time, phaco
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Victus Group (Experimental): The anterior capsulotomy and lens fragmentation will be performed by means of femtosecond laser surgery
  Interventions: Device: Victus
- Conventional Group (Other): The Conventional Group acts as a control group where the capsulotomy as well as the lens fragmentation is performed manually
  Interventions: Device: Conventional Phaco

INTERVENTIONS:
Device: Victus — The anterior capsulotomy and lens fragmentation will be performed by means of femtosecond laser surgery
  Arms: Victus Group
Device: Conventional Phaco — The capsulotomy as well as the lens fragmentation is performed manually.
  Arms: Conventional Group

SUMMARY:
Cataract surgery is among the world's most frequently performed operations. It involves removal of an opaque lens from the human eye and implantation of an artificial lens. The operation is performed under local anaesthesia using ultrasound technology, by which the lens is emulsified and removed by suction.

Femtosecond laser-assisted cataract surgery is a new innovative surgical procedure that can improve the quality of cataract surgery and provide a new best possible standard of quality. In contrast to the conventional method the capsulotomy and the fragemntation are fully automatically performed with a femtosecond laser. In addition, the lens is fragmented by the laser, which substantially facilitates its removal and reduces the operation time.

Study to investigate whether the femtosecond laser cataract surgery causes any significant differences in clinical outcomes as compared to the conventional, manual continuous curvilinear capsulorhexis (CCC).

Effective phako time (EPT) is defined as duration of phakoemulsifikation of the crystalline lens.

EPT of conventional surgery at intraoperative visit > EPT oflaser-assisted surgery at intraoperative visit

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* related cataract
* Ability to follow instructions from the treatment team
* Both eyes to receive surgery

Exclusion Criteria:

* Narrow pupils (in ther. mydriasis <6mm)
* Narrow orbits
* Sunken eyes
* manifest glaucoma treated with anti-glaucomatous therapy or prior surgery
* Conditions that pose a high risk of complications during surgery
* Known sensitivity to planned concomitant medications
* Patients with disorders of the ocular muscle, such as nystagmus or strabismus
* Patients who are blind on one eye
* Acute or chronic systemic and/or ocular illnesses that are clinically significant and will increase the risk to the subject or confound the outcomes of this study, such as but not restricted to diabetes mellitus, autoimmune/rheumatic or connective tissue diseases, dementia or epilepsy.
* Patients who are pregnant or nursing
* Patients who do not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Effective Phaco Time | surgery day
  EPT of the conventional cataract surgery (mesured intraoperativ = Visit 2) is smaller or equal to the EPT of the Laser-assisted cataract surgery (meausred intraoperativ = Visit 2)

SECONDARY OUTCOMES:
IOL overlap | 1 month, 3 and 6 months
  The difference in the IOL overlap between group A and B. The IOL overlap, ΔROverlap, is the euclidian distance between the center of mass of the capsulotomy and the center of mass of the IOL, representing the symmetry of the IOL-Capsulotomy aperture- overlap
IOL Centration | 1 month, 3 and 6 months
  The difference in the IOL centration between group A and B. The IOL centration is the euclidian distance between the center of mass of the IOL and the center of mass of the dilated pupil

OTHER OUTCOMES:
patients subjective perception | 1 day
  Patients' subjective perceptions of the two operative procedures
cornea, retina | 1 month, 3 and 6 month
  Effects of the surgical techniques on the cornea and retina as assessed by optical coherence tomography, endothelial cell count or Pentacam.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, MD, Principal Investigator — AKh Linz, Ophthalmology
Locations (1):
- AKh Linz, Linz, Upper Austria, Austria